CLINICAL TRIAL: NCT01814514
Title: Early Intra Ocular- Pressure Control Using Aqueous Suppressive Agents After Ahmed Glaucoma Valve Implantation
Brief Title: Safety Study of Aqueous Suppression After Ahmed Glaucoma Valve (AGV) Implantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zahra Rabbani Khah (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Zahra Rabbani Khah, ophthalmologist, Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90166
Record Dates: First submitted 2013-03-07; First posted 2013-03-20 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Hypertensive Phase
Keywords: hypertensive; phase; success rate; AGV
MeSH Terms: interventions — dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Timolol-trusopt (Active Comparator): Dosage:One drop/12hours,duration:3 months
  Interventions: Drug: Timolol-trusopt
- placebo,Artificial tear (Placebo Comparator): dosage:one drop/12 hours,duration:3 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Timolol-trusopt
  Other Names: cosopt
  Arms: Timolol-trusopt
Drug: placebo
  Arms: placebo,Artificial tear

SUMMARY:
The AGV implant is designed to open when the IOP is between 8 mmHg and 10 mmHg, and thus maintains an IOP of 8 mmHg or higher. In the early period after glaucoma drainage device (GDD) surgery the intraocular pressure (IOP) classically goes through 2 phases. The hypotensive phase occurs immediately after surgery, lasts around 1 week. This is followed by the hypertensive period where the IOP tends to rise steadily above 21mmhg.

The hypertensive response seems to occur more commonly after Ahmed GDD surgery than nonvalved implants, It was reported to occur in 40% to 80% of cases. Although the hypertensive phase can last as long as 6 months it is usually during the first 1 to 4 weeks, when there is intense congestion of the bleb wall, that IOP is highest.

Previous study showed that when aqueous comes into contact with conjunctiva and Tenon's capsule,an inflammatory reaction occurs.Factors such as prostaglandins, eicosanoids, tissue growth factor beta (TGF β)has been shown to occur in glaucomatous aqueous. These mediators induce an inflammatory reaction, and if excessive, will result in fibrosis and poor functioning of the bleb. High pressure within the bleb also results in the secretion of TGF β by the bleb lining. It may result in inflammation of the bleb wall and subsequent fibrosis and poor bleb function. The investigators supposed that with early use of aqueous suppressant medication after AGV implantation, the concentration of inflammatory mediators decreased in subconjunctival space and may lead to better IOP control after shunt surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with uncontrolled glaucoma requiring AGV device implantation.

Exclusion Criteria:

1. History of AGV implantation
2. Allergy to Anti glaucoma medication
3. unable to come for follow up
4. Known contraindication to beta blacker such as asthma- chronic obstructive pulmonary disease (COPD). Heart failure heart block
5. Learning difficulty- mental illness or severely ill

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure-hypertensive phase success rate | during first 3 months
  during first 3 months

SECONDARY OUTCOMES:
intraocular pressure success rate | after 12 months
  after 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Labbafinejad medical center, Tehran, Iran